CLINICAL TRIAL: NCT05822271
Title: Evaluation of Surgical Outcomes of Patients Treated With the Surgery First Approach and Aligners
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rio de Janeiro State University (Other)
Responsible Party: Principal Investigator, Arthur Cunha, Clinical Professor, Rio de Janeiro State University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 51444621.0.0000.5259
Record Dates: First submitted 2023-03-31; First posted 2023-04-20 (Actual); Last update posted 2024-12-02 (Actual); Status verified 2024-11

CONDITIONS: Malocclusion, Angle Class III
Keywords: Surgery-First; Orthognathic; Aligner; Aesthetic Treatment
MeSH Terms: conditions — Malocclusion, Angle Class III | interventions — Orthognathic Surgery

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Orthodontic Aligner treatment (Experimental)
  Interventions: Procedure: Orthognathic Surgery
- Orthodontic fixed appliance treatment (Active Comparator)
  Interventions: Procedure: Orthognathic Surgery

INTERVENTIONS:
Procedure: Orthognathic Surgery — Type of surgery performed to correct skeletal malocclusions

SUMMARY:
The purpose of this prospective study is to compare treatment outcomes and the quality of life of skeletal Class III patients treated with conventional fixed appliances and aligners undergoing Surgery-first approach. Data will be collected through validated questionnaires: OQLQ (Orthognathic Quality of Life Questionnaire), OHIP-14 (Oral Health Impact Proﬁle), SF-36 (Medical Outcomes Study 36 - Item Short-Form Health Survey) and IOTN (Index of Orthodontic Treatment Need).

ELIGIBILITY:
Inclusion Criteria:

* Adults;
* Skeletal malocclusion;
* ANB Angle zero or negative;
* Witts negative;
* Etiology: mandibular excess, a maxillary deficiency, or a combination of both;
* Indication for bimaxillary surgery;

Exclusion Criteria:

* Previous orthodontic treatment;
* Craniofacial anomaly or previous fracture of the facial bones;
* Total edentulism;
* Deep curve of Spee;
* Vertical asymmetry;
* Any medication use that contraindicates surgical treatment.

Ages: 17 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-01-30 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Quality of life accessed by validated questionnaires. | at the end of orthodontic treatment (up to 2 years).
  Comparison between quality of life changes in the two groups at the end of treatment.

SECONDARY OUTCOMES:
Periodontal status. | at the end of orthodontic treatment (up to 2 years).
  Comparison between periodontal changes in the two groups at the end of the treatment.
Treatment duration. | at the end of orthodontic treatment (up to 2 years).
  Comparison between treatment time in the two groups at the end of the treatment.
Facial changes as measured by tomographic superimposition of the face. | at the end of orthodontic treatment (up to 2 years).
  Comparison between facial changes in the two groups at the end of the treatment.
Incisors inclination | at the end of orthodontic treatment (up to 2 years).
  Quantitative assessment of incisors inclination between the two groups as measured by tomographic superimposition at the end of orthodontic treatment.
Alveolar bone changes around incisors. | at the end of orthodontic treatment (up to 2 years).
  Comparison between the alveolar bone changes around incisors by tomographic.
Swelling as measured by tomographic images. | 12 months post-operative.
  Comparison between facial swelling in the two groups after orthognathic surgery.
Surgery stability as measured by tomographic superimposition. | 12 months post-operative.
  Comparison between surgery stability in the two groups at the end of the treatment.
Changes in relationship between maxilla and mandible as measured by tomographic superimposition of the cranial base. | 12 months post-operative.
  Comparison between the changes of the relationship among maxilla and mandible in the two groups at the end of the treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Rio de Janeiro State University, Rio de Janeiro, Brazil

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Miguel JA, Palomares NB, Feu D. Life-quality of orthognathic surgery patients: the search for an integral diagnosis. Dental Press J Orthod. 2014 Jan-Feb;19(1):123-37. doi: 10.1590/2176-9451.19.1.123-137.sar. PMID 24713569
- [Background] Palomares NB, Celeste RK, Miguel JA. Impact of orthosurgical treatment phases on oral health-related quality of life. Am J Orthod Dentofacial Orthop. 2016 Feb;149(2):171-81. doi: 10.1016/j.ajodo.2015.07.032. PMID 26827973
- [Background] Baek SH, Ahn HW, Kwon YH, Choi JY. Surgery-first approach in skeletal class III malocclusion treated with 2-jaw surgery: evaluation of surgical movement and postoperative orthodontic treatment. J Craniofac Surg. 2010 Mar;21(2):332-8. doi: 10.1097/SCS.0b013e3181cf5fd4. PMID 20186090
- [Background] Peiro-Guijarro MA, Guijarro-Martinez R, Hernandez-Alfaro F. Surgery first in orthognathic surgery: A systematic review of the literature. Am J Orthod Dentofacial Orthop. 2016 Apr;149(4):448-62. doi: 10.1016/j.ajodo.2015.09.022. PMID 27021449
- [Background] Feu D, de Oliveira BH, Palomares NB, Celeste RK, Miguel JAM. Oral health-related quality of life changes in patients with severe Class III malocclusion treated with the 2-jaw surgery-first approach. Am J Orthod Dentofacial Orthop. 2017 Jun;151(6):1048-1057. doi: 10.1016/j.ajodo.2016.10.034. PMID 28554450
- [Background] Flores-Mir C, Brandelli J, Pacheco-Pereira C. Patient satisfaction and quality of life status after 2 treatment modalities: Invisalign and conventional fixed appliances. Am J Orthod Dentofacial Orthop. 2018 Nov;154(5):639-644. doi: 10.1016/j.ajodo.2018.01.013. PMID 30384934
- [Background] Buschang PH, Shaw SG, Ross M, Crosby D, Campbell PM. Comparative time efficiency of aligner therapy and conventional edgewise braces. Angle Orthod. 2014 May;84(3):391-6. doi: 10.2319/062113-466. Epub 2013 Nov 18. PMID 24749702
- [Background] Miller KB, McGorray SP, Womack R, Quintero JC, Perelmuter M, Gibson J, Dolan TA, Wheeler TT. A comparison of treatment impacts between Invisalign aligner and fixed appliance therapy during the first week of treatment. Am J Orthod Dentofacial Orthop. 2007 Mar;131(3):302.e1-9. doi: 10.1016/j.ajodo.2006.05.031. PMID 17346581
- [Background] Liou EJ, Chen PH, Wang YC, Yu CC, Huang CS, Chen YR. Surgery-first accelerated orthognathic surgery: orthodontic guidelines and setup for model surgery. J Oral Maxillofac Surg. 2011 Mar;69(3):771-80. doi: 10.1016/j.joms.2010.11.011. Epub 2011 Jan 22. PMID 21257249
- [Background] Villegas C, Uribe F, Sugawara J, Nanda R. Expedited correction of significant dentofacial asymmetry using a "surgery first" approach. J Clin Orthod. 2010 Feb;44(2):97-103; quiz 105. No abstract available. PMID 20552809
- [Background] Liao YF, Chen YA, Chen YC, Chen YR. Outcomes of conventional versus virtual surgical planning of orthognathic surgery using surgery-first approach for class III asymmetry. Clin Oral Investig. 2020 Apr;24(4):1509-1516. doi: 10.1007/s00784-020-03241-4. Epub 2020 Feb 25. PMID 32100114
- [Background] Liao YF, Lo SH. Surgical Occlusion Setup in Correction of Skeletal Class III Deformity Using Surgery-First Approach: Guidelines, Characteristics and Accuracy. Sci Rep. 2018 Aug 3;8(1):11673. doi: 10.1038/s41598-018-30124-2. PMID 30076359
- [Background] de Leyva P, Eslava JM, Hernandez-Alfaro F, Acero J. Orthognathic surgery and aligners. A comparative assessment of periodontal health and quality of life in postsurgical orthodontic treatment with aligners versus traditional fixed appliances: a randomized controlled trial. Med Oral Patol Oral Cir Bucal. 2023 May 1;28(3):e208-e216. doi: 10.4317/medoral.25555. PMID 37026606
- [Derived] Cunha A, Silva LKA, da Silveira HM, Miguel JAM. Impact on Oral Health-Related Quality of Life in Skeletal Class III Patients Treated With Orthognathic Surgery-First Approach Using Orthodontic Aligners or Fixed Appliances: A Controlled Clinical Study. Orthod Craniofac Res. 2026 Feb;29(1):112-121. doi: 10.1111/ocr.70054. Epub 2025 Nov 7. PMID 41200809